CLINICAL TRIAL: NCT04461613
Title: Developing and Testing Instrument to Measure Physical Activity in Charcot-Marie-Tooth: a Pilot Project
Brief Title: Physical Activity in Persons With Charcot-Marie-Tooth: Developing a Measurement Instrument
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian National Advisory Unit on Rare Disorders (NKSD) (Unknown); University of Oslo (Other); Foreningen for Muskelsyke (Unknown)
Responsible Party: Principal Investigator, Kristin Ørstavik, Consultant in Neurology and Head of Section for Rare Neuromuscular disorders including EMAN, Department of Neurology, Oslo University Hospital, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2020/94587
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hereditary Motor and Sensory Neuropathy; Charcot-Marie-Tooth; Polyneuropathies
Keywords: CMT; IPAQ; NMD; Charcot-Marie-Tooth; International Physical Activity Questionnaire; neuromuscular disorders; activity diary; hereditary neuropathy
MeSH Terms: conditions — Hereditary Sensory and Motor Neuropathy; Charcot-Marie-Tooth Disease; Polyneuropathies; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Two groups of people with CMT will compare an original International Physical Activity Questionnaire short form (IPAQ-sf) and a revised one with a 7-days physical activity diary. The first group will begin with the original version and end with a revised one. The second group will begin with a revised IPAQ-sf and end with the original one. Both groups will also need to complete a 7-days activity diary two times.
Who Masked: Care Provider, Investigator
Masking Description: Study participants will receive an unmarked envelope consisting of all study material. The order of the study questionnaires inside the unmarked envelope will be randomized and sealed by the first researcher. The first researcher will give them to the second researcher who will again shuffle the envelopes order (without the first researcher present) before giving them to the care provider. The care provider will give the study envelope to the study participants. Therefore, investigators and care provider will be masked to the contents of the unmarked study envelope and cannot selectively assign the participants to a certain group. However, the study participants might recognize the original IPAQ if she/he received this questionnaire in the past.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In the first week, this group will receive a physical activity diary and be required to fill it out for 7 days. After completion of the activity diary, group 1 will receive an original International Physical Activity Questionnaire short form (IPAQ-sf). Group 1 will be asked to fill it out with information about physical activities in the last 7 days.
  In the second week, the group will need to fill another physical activity diary for 7 days. After the completion of this, group 1 will be asked to fill a revised version of IPAQ-sf to describe physical activities in the last 7 days.
  Interventions: Other: Original IPAQ followed by a revised one.
- Group 2 (Experimental): In the first week, this group will receive a physical activity diary and be required to fill it out for 7 days. After completion of the activity diary, group 2 will receive a revised version of International Physical Activity Questionnaire short form (IPAQ-sf). Group 2 will be asked to fill it out with information about physical activities in the last 7 days.
  In the second week, the group will need to fill another physical activity diary for 7 days. After the completion of this, group 2 will be asked to fill an original IPAQ-sf to describe physical activities in the last 7 days.
  Interventions: Other: Revised IPAQ followed by an original one.

INTERVENTIONS:
Other: Original IPAQ followed by a revised one. — Comparing two questionnaires (a revised version and an original International Physical Activity Questionnaire short form) with an activity diary.
  Arms: Group 1
Other: Revised IPAQ followed by an original one. — Comparing two questionnaires (a revised version and an original International Physical Activity Questionnaire short form) with an activity diary.
  Arms: Group 2

SUMMARY:
The project will develop knowledge about physical activity in persons with Charcot-Marie-Tooth (CMT) in Norway. We plan to explore instruments to measure physical activity level for the target-group at the community level. We want to understand which type of activities, activity intensities and how persons with CMT perform habitual physical activity. Subsequently, a physical activity measurement instrument adapted to persons with CMT will be developed. This instrument can be used in a future intervention project to promote physical activity in this group.

DETAILED DESCRIPTION:
Charcot-Marie-Tooth (CMT) is a condition that potentially affects daily life function including physical activity. Currently, there is no specific treatment. To prevent physical deconditioning, physical activity recommended. Furthermore, other studies have found the benefit of being physically active, including people with neuromuscular disorders (NMD). .

Apart from the physical activity in a rehabilitation center, physical activity also needs to be maintained at the community level in people's everyday life. To measure physical activity level in the community, we need an instrument that is designed for doing so. A questionnaire can be used to collect information about type of activity, activity duration and intensity. The instruments available so far to measure physical activity at the community level are not specifically adapted to persons with CMT. Therefore, this study will focus on revising the questionnaire based on the inputs from persons with CMT themselves. Furthermore, the revised questionnaire will be compared with the original one in addition to yet another instrument.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a genetically confirmed CMT diagnosis.
* Residing in Norway
* Age between 18 to 65 years old.

Exclusion Criteria:

* Had major surgery within three months prior to the study period.
* Experiencing serious illness (e.g. bedridden, hospitalized).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Total physical activity duration | 16 days
  Correlations of the total physical activity duration measured using original and revised International Physical Activity Questionnaire short form (IPAQ-sf) with an activity diary (in minutes/week).
  The original IPAQ-sf has been used in Norwegian context and available in Norwegian language. It has a criterion validity of 0.30 (95% CI 0.23-0.36) against accelerometer count and 0.30-0.46 for correlation with a physical activity diary physical activity level (in MET minutes/week). The content of the revised IPAQ-sf was formulated based on the inputs from experts, including the persons with CMT themselves in our reference group. The revised IPAQ-sf will be compared with the original IPAQ-sf in this pilot project.

SECONDARY OUTCOMES:
Physical activity duration for different intensities from original and revised IPAQ-sf | 16 days
  Correlations of the physical activity duration at three different intensities: high/vigorous, moderate, and light/walking, measured using original and revised IPAQ-sf with an activity diary (in minutes/week).
  Both original and revised IPAQ-sf can provide description of physical activity level in three different intensities: high/vigorous, moderate, and light/walking. In the activity diary, the Borg's scale will be used to describe intensity in categories: high, moderate, and light. The Borg's scale has weighted mean validity coefficients 0.57-0.72 for various physiological measurements, including: heart rate, blood lactate, %VO2max, VO2, ventilation, and respiration rate.
Qualitative inputs from the pilot study participants for all of the study instruments | 16 days
  Inputs and comments from pilot study participants for the original IPAQ-sf, revised IPAQ-sf, and activity diary.
  In this pilot project, we provided field for comments for each point of question in all three questionnaires: original IPAQ-sf, revised IPAQ-sf, and physical activity diary. These qualitative inputs will be analysed for further development and improvement of the study instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ørstavik, MD, Ph.D., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No